CLINICAL TRIAL: NCT03921918
Title: Evaluation of Fluid-Filled Expression Core Technology Study - I
Acronym: Effect-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medela AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MHM1801
Record Dates: First submitted 2019-04-11; First posted 2019-04-19 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2019-11

CONDITIONS: Breast Pumping
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of Fluid Expression Technology (Other): This study aims to provide important insights with respect to the safety, performance, and real-life usability of pumping technology
  Interventions: Device: Breast Pump

INTERVENTIONS:
Device: Breast Pump — Hydraulic Breast pump

SUMMARY:
A functional model of a fluid-filled, smaller dead volume breast pump has been developed in order to more closely mimic the breastfeeding infant. The technology of fluid-filled pumping has been tested in one prior clinical study and has now progressed to a complete prototype with which the user can assemble, pump, disassemble, clean and reuse.

DETAILED DESCRIPTION:
Current breast pumps function in a way that is different to breastfeeding. These include the seal to the breast, the movement of the nipple, the sensations of warmth and moisture, the variability in frequency, and the strength of the applied vacuum. During breastfeeding the mother's nipple and the infant's mouth form a chamber that is a fluid-filled, no dead volume system, which is needed to create a working vacuum to remove milk from the breast. There is no air visible in the natural system according to ultrasound measurements. This is unlike breast pumps which use an air-filled, large dead volume system, to create a working vacuum. Therefore, a functional model of a fluid-filled, smaller dead volume breast pump has been developed in order to more closely mimic the breastfeeding infant. The technology of fluid-filled pumping has been tested in one prior clinical study and has now progressed to a complete prototype with which the user can assemble, pump, disassemble, clean and reuse.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥ 18 years old
2. Infant is ≥1 and ≤6 month old
3. Subject and baby are healthy according to self-declaration in the "Mother and infant health questionnaire"
4. Subject is predominantly breastfeeding (80% of all feeds, i.e. ≤150 ml formula/day or equal representative amount of solid food)
5. The subject agrees to pump or feed the last time a minimum of 2 hours (hr) before the start of the pumping session at the study site
6. The subject agrees to photographs/3 D scan of the breast and upper body (no face),
7. The subject agrees to a video while pumping
8. The subject signs the informed consent documentation
9. Subject agrees that a maximum of 2 male team members can be present in the room to conduct the usability part of the study
10. The mother accepts that the pumped milk in visit 2 must be donated to the study i.e. cannot be fed to the baby

Exclusion Criteria:

1. The subject has a nipple size ≥ 21 mm
2. Mastitis (any breast within two weeks prior to enrolment)
3. Engorgement (any breast within two weeks prior to enrolment).
4. Case of current infection as self-declared in the Mother and infant health questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 26 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Recording all Adverse Events | 3 months
  Recording all AE and evaluating the (time of) occurrence, type, seriousness, expectedness, relatedness, and outcome of the adverse events
Observing pump performance | 3 months
  Measuring milk flow volume including time to first ejection.

SECONDARY OUTCOMES:
Measureing user acceptance | 3 months
  Analysing the User Experience Questionnaire as per Laugwitz, Held & Schrepp (2017)

CONTACTS AND LOCATIONS:
Overall Officials: Beatrix Mascher, MBA, Principal Investigator — Clinical Affairs within Medical Reseach and R&D
Locations (1):
- Medela AG, Baar, Switzerland

IPD SHARING:
Plan to Share IPD: No